CLINICAL TRIAL: NCT03933826
Title: CISTO: Comparison of Intravesical Therapy and Surgery as Treatment Options for Bladder Cancer
Acronym: CISTO
Status: Active, not recruiting | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, John Gore, Associate Professor, School of Medicine: Urology, University of Washington
Other Study IDs: SITE00001017; PCS-2017C3-9380 (Other: PCORI); RG1121143 (Other: Fred Hutch/University of Washington Cancer Consortium); NCI-2020-06082 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-04-19; First posted 2019-05-01 (Actual); Results first posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Bladder Cancer; Cancer of the Bladder, Recurrent; Non-muscle Invasive Bladder Cancer
Keywords: pragmatic trial; Bacillus Calmette-Guerin (BCG); urinary bladder neoplasms; urogenital neoplasms; radical cystectomy; neoplasms by site; neoplasms; urinary bladder disease; immunologic factors; caregivers; physiological effects of drugs; immunologic adjuvants; urologic diseases
MeSH Terms: conditions — Urinary Bladder Neoplasms; Recurrence; Non-Muscle Invasive Bladder Neoplasms; Urogenital Neoplasms; Neoplasms by Site; Neoplasms; Urinary Bladder Diseases; Urologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients who have selected radical cystectomy: Patients with a diagnosis of recurrent high-grade NMIBC who have selected radical cystectomy
- Patients who have selected bladder-sparing therapy: Patients with a diagnosis of recurrent high-grade NMIBC who have selected bladder-sparing therapy (BST)

SUMMARY:
Bladder cancer is the most common urinary tract cancer and the 5th most common cancer in the US (1). Yet bladder cancer research is underfunded relative to other common cancers. As a result, bladder cancer care is prone to evidence gaps that produce decision uncertainty for both patients and clinicians. The Comparison of Intravesical Therapy and Surgery as Treatment Options (CISTO) for Bladder Cancer Study has the potential to fill these critical evidence gaps, change care pathways for the management of non-muscle-invasive bladder cancer (NMIBC), and provide for personalized, patient-centered care. The purpose of CISTO is to conduct a large prospective study that directly compares the impact of medical management versus bladder removal in recurrent high-grade NMIBC patients with Bacillus Calmette-Guerin (BCG) failure on clinical outcomes and patient and caregiver experience using standardized patient-reported outcomes (PROs).

DETAILED DESCRIPTION:
Most bladder cancer patients (74%) present with NMIBC where the cancer is limited to the lining or support layer of the bladder. High-grade NMIBC is treated initially with endoscopic resection and intravesical immunotherapy, followed by bladder instillations of BCG. Most patients with high-risk, high-grade NMIBC are able to retain their bladders and avoid more invasive treatments. However, 24-61% of patients will have their cancers recur within 12 months of treatment with BCG (BCG failures), and they have limited treatment options. National guidelines recommend consideration between two alternatives: additional medical management and radical cystectomy (removal of the bladder). Selecting between these options involves weighing the risk of progression of bladder cancer and loss of a window of potential cure versus the risk of morbidity and loss of quality of life (QOL) with bladder removal. This complex decision-making engages patients and their caregivers, who may be impacted by the urinary, sexual, and bowel dysfunctions that can occur with NMIBC treatment.

The investigators will evaluate this research question on a large scale in real world practice settings including academic and community-based practices and examine patient-centered outcomes. The investigators have engaged stakeholders with diverse perspectives relevant to this research question, including patients, caregivers, national patient advocacy organizations, national medical specialty organizations, guideline developers, health care payers, and industry. By engaging broad expertise relevant to this research question, the investigators will ensure that the study results will help NMIBC patients whose cancer recurs after BCG treatment make more informed decisions that improve the health outcomes that are important to them.

CISTO is an observational study that will not affect the treatment that patients chose. Patient surveys will occur at study entry and at follow-up assessments for up to four years. There will also be a qualitative sub-study that will include interviews of approximately 50 patients and 25 caregivers recruited from the observational cohort study.

ELIGIBILITY:
Patient Eligibility, Inclusion Criteria:

1. Adult 18 years of age or older; and
2. Presenting with high-grade NMIBC established by anatomic pathology as tumor stage classification Tis, Ta, or T1, and with:

   1. Pathology documentation from any hospital/clinic/medical center, and
   2. More than 50% urothelial carcinoma component in the specimen
3. History of high-grade NMIBC established by anatomic pathology as tumor stage classification Tis, Ta, or T1; and
4. Attempted or received induction BCG (at least 3 out of 6 instillations) at any point in time; and
5. In the previous 12 months, received at least one instillation of any intravesical agent (induction or maintenance) or one administration of systemic therapy for NMIBC treatment.

Patient Eligibility, Exclusion Criteria:

1. Any plasmacytoid or small cell (neuroendocrine) component in the pathology (past or current presentation);
2. Previous history of cystectomy or radiation therapy for bladder cancer;
3. Previous history of muscle-invasive bladder cancer or metastatic bladder cancer;
4. Any history of upper tract urothelial carcinoma;
5. Incarcerated in a detention facility or in police custody (patients wearing a monitoring device can be enrolled) at baseline/screening;
6. Contraindication to radical cystectomy (e.g., American Society of Anesthesiologists (ASA) physical status of 4, patient not considered a radical cystectomy candidate due to comorbidity);
7. Contraindication to medical therapy (i.e., intolerant of all medical therapies);
8. Unable to provide written informed consent in English;
9. Unable to be contacted for research surveys;
10. Planning to participate in a Phase I or Phase II interventional clinical trial for NMIBC (unless in the control/comparator arm of a Phase II trial) or any blinded interventional trial for NMIBC.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of recurrent high-grade NMIBC who are considering second-line treatment will be approached for participation in this observational study in addition to their caregivers. Enrollment at each site will aim for a 2:1 ratio of participants selecting bladder-sparing therapy to radical cystectomy in order to ensure adequate enrollment of radical cystectomy patients. There will also be a qualitative sub-study that will include interviews of 50 patients and 25 caregivers recruited from the observational cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 570 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2029-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John L Gore, MD, Principal Investigator — University of Washington
Locations (36):
- United States (36):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Cancer Center, Phoenix, Arizona
  - USC/Norris Comprehensive CA Center, Los Angeles, California
  - UCLA, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - LSU Healthcare Network - Multi Specialty Clinic, Metairie, Louisiana
  - Johns Hopkins University, School of Medicine, Baltimore, Maryland
  - Chesapeake Urology Research Associates, Hanover, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Michigan Medicine Rogel Cancer Center, Ann Arbor, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Comprehensive Urology -- A Division of Michigan Healthcare Professionals, Royal Oak, Michigan
  - Albert Einstein College of Medicine, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Asante Rogue Regional Medical Center, Medford, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Carolina Urologic Research Center, LLC, Myrtle Beach, South Carolina
  - Urology Associates, P.C., Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified study data will be shared according to the PCORI policy for data management and data sharing.
Supporting Information: Study Protocol, SAP
Time Frame: The PCORI-designated repository will make the data available for third-party requests when PCORI makes the Final Research Report available on the PCORI website pursuant to PCORI's Process for Peer Review of Primary Research and Public Release of Research Findings. Data will be available in perpetuity.
Access Criteria: Individual investigators or teams of investigators seeking access to data from PCORI-funded studies must complete and submit a data request form to the PCORI-designated repository.

REFERENCES:
- [Derived] Gore JL, Wolff EM, Nash MG, Comstock BA, Gilbert SM, Chang SS, Chisolm S, MacLean DB, Wright JL, Kates MR, Pohar KS, Guzzo TJ, Bivalacqua TJ, Nepple KG, Montgomery JS, Scarpato KR, Woldu SL, Master VA, Chen DYT, Mossanen M, Daneshmand S, O'Neil BB, Tyson MD, Westerman ME, Kamat AM, Mansour AM, Chamie K, Riggs SB, Kukreja JB, Modi PK, Garg T, Peyton CC, Nix JW, Dickstein R, Gadzinski AJ, Sankin A, Shore ND, Lane BR, Bassett JC, Patel S, Morris DS, Macleod LC, Lee EK, Ritch CR, Follmer KM, Lee JR, Kim SM, Kessler LG, Smith AB; CISTO Collaborative group. Twelve-Month Results From the CISTO Study Comparing Radical Cystectomy Versus Bladder-Sparing Therapy for Recurrent High-Grade Non-Muscle-Invasive Bladder Cancer. J Clin Oncol. 2026 Feb;44(4):274-285. doi: 10.1200/JCO-25-01324. Epub 2025 Dec 15. PMID 41397208
- [Derived] Gore JL, Wolff EM, Comstock BA, Follmer KM, Nash MG, Basu A, Chisolm S, MacLean DB, Lee JR, Lotan Y, Porten SP, Steinberg GD, Chang SS, Gilbert SM, Kessler LG, Smith AB; CISTO Collaborative. Protocol of the Comparison of Intravesical Therapy and Surgery as Treatment Options (CISTO) study: a pragmatic, prospective multicenter observational cohort study of recurrent high-grade non-muscle invasive bladder cancer. BMC Cancer. 2023 Nov 18;23(1):1127. doi: 10.1186/s12885-023-11605-8. PMID 37980511

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients who have selected bladder-sparing therapy | Patients who have selected radical cystectomy
Started | 371 | 199
12-months from enrollment | 303 | 174
Completed | 303 | 174
Not Completed | 68 | 25
Not completed — Withdrawal by Subject | 8 | 1
Not completed — Death | 19 | 11
Not completed — Lost to Follow-up | 41 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients who have selected bladder-sparing therapy | Patients who have selected radical cystectomy | Total
Number analyzed (Participants) | 371 | 199 | 570
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.4 (8.3) | 69.6 (9.1) | 71.4 (8.7)
Age, Customized [Count of Participants; unit: Participants] — Categorical age with cut off of 75 years
  Participants
    greater than or equal to 75 years | 150 | 62 | 212
    Less than 75 years | 221 | 137 | 358
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 39 | 117
  Male | 293 | 160 | 453
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 17 | 56
  Not Hispanic or Latino | 332 | 182 | 514
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 8 | 26
  White | 341 | 184 | 525
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 4 | 2 | 6
Partner status [Count of Participants; unit: Participants] — Has a spouse or partner (partnered) or unpartnered
  Participants
    Partnered | 288 | 170 | 458
    Unpartnered | 83 | 29 | 112

OUTCOME MEASURES:

1. Primary Outcome: Patient-reported Quality of Life as Measured by the Physical Function Scale of the European Organization for Research and Treatment of Cancer Quality-of-Life-Questionnaire-Core-30 (EORTC QLQ-C30)
Description: The primary outcome of patient-reported quality of life is measured by the EORTC QLQ-C30 Physical Function scale. The scale ranges in score from 0 to 100, with higher function scores indicating better health. Scale score is calculated by transforming individual item scores into a 0 to 1 scale, taking the mean, and multiplying by 100. Each scale requires responses for at least 50% of the items in order to be calculated.
Time Frame: 12 months after enrollment
Population: We performed tenfold multiple imputation (MICE R package) for all missing outcomes and covariates for analyses of all patient-reported outcomes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients who have selected bladder-sparing therapy | Patients who have selected radical cystectomy
Number analyzed (Participants) | 304 | 174
score on a scale | 85.0 (18.9) | 86.5 (17.5)
Statistical Analysis 1: Comparison: Patients who have selected bladder-sparing therapy vs Patients who have selected radical cystectomy; Test type: Superiority; p < 0.05, TMLE — We tested the hypothesis that the average treatment effect (ATE) is different from zero. This was the only hypothesis test in our primary manuscript, and so no adjustment for multiple comparisons is necessary; TMLE stands for targeted maximum likelihood estimation; Average treatment estimate (ATE) = 0.9, 95% CI 2-sided [-0.6 to 2.4] — The causal mean difference in outcomes if all patients had been treated with radical cystectomy versus with bladder-sparing therapy. A positive value indicates greater physical functioning associated with radical cystectomy

2. Primary Outcome: Patient-reported Quality of Life as Measured by the Physical Function Scale of the European Organization for Research and Treatment of Cancer Quality-of-Life-Questionnaire-Core-30 (EORTC QLQ-C30)
Description: Patient-reported quality of life is measured by the EORTC QLQ-C30 Physical Function scale. The scale ranges in score from 0 to 100, with higher function scores indicating better health. Scale score is calculated by transforming individual item scores into a 0 to 1 scale, taking the mean, and multiplying by 100. Each scale requires responses for at least 50% of the items in order to be calculated.
Time Frame: 24 months after enrollment
Reporting Status: Not Posted

3. Primary Outcome: Patient-reported Quality of Life as Measured by the Physical Function Scale of the European Organization for Research and Treatment of Cancer Quality-of-Life-Questionnaire-Core-30 (EORTC QLQ-C30)
Description: as for outcome 2
Time Frame: 60 months after enrollment
Reporting Status: Not Posted

4. Secondary Outcome: Patient Self-reported Urinary Health as Measured by the Bladder Cancer Index Urinary Summary Score
Description: The evaluation of the effect of treatment choice on patient-reported urinary health, as measured by the Bladder Cancer Index (BCI). The BCI consists of 36 items, with 4- or 5-point Likert response scales, covering 3 primary domains: urinary, bowel, and sexual. For each domain a summary score is constructed from the items used to calculate the two subscale scores (function and bother). Scores are calculated by transforming item responses into a 0 to 100 scale and calculating the mean of the standardized items. Higher scores indicate better health status. To calculate a score, a minimum of 80% completed items is required.
Time Frame: 12 months after enrollment
Population: We imputed missing outcomes and covariates for TMLE analyses of this outcome. Therefore, all participants who enrolled in CISTO are included whether or not they completed that outcome. The mean and standard deviation for this outcome was calculated using only participants who completed this outcome (n = 292 and 166 for bladder-sparing therapy and radical cystectomy arms, respectively).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients who have selected bladder-sparing therapy | Patients who have selected radical cystectomy
Number analyzed (Participants) | 292 | 166
score on a scale | 85.3 (16.7) | 83.8 (14.2)
Statistical Analysis 1: Comparison: Patients who have selected bladder-sparing therapy vs Patients who have selected radical cystectomy; Test type: Other — We did not conduct a hypothesis test for this outcome. We presented an estimate of the average treatment effect (ATE); TMLE = 1.2, 95% CI 2-sided [-0.5 to 2.9] — The ATE is interpreted as the causal mean difference in outcomes if all patients had been treated with RC versus having been treated with BST. A positive value indicates greater urinary health associated with radical cystectomy

5. Secondary Outcome: Patient Self-reported Urinary Health as Measured by the Bladder Cancer Index Urinary Summary Score
Description: as for outcome 4
Time Frame: 24 months after enrollment
Reporting Status: Not Posted

6. Secondary Outcome: Patient Self-reported Urinary Health as Measured by the Bladder Cancer Index Urinary Summary Score
Description: as for outcome 4
Time Frame: 60 months after enrollment
Reporting Status: Not Posted

7. Secondary Outcome: Patient Self-reported Sexual Health as Measured by the Bladder Cancer Index Sexual Summary Score
Description: The evaluation of the effect of treatment choice on patient-reported sexual health, as measured by the Bladder Cancer Index (BCI). The BCI consists of 36 items, with 4- or 5-point Likert response scales, covering 3 primary domains: urinary, bowel, and sexual. For each domain a summary score is constructed from the items used to calculate two subscale scores (function and bother). Scores are calculated by transforming item responses into a 0 to 100 scale and calculating the mean of the standardized items. Higher scores indicate better health status. To calculate a score, a minimum of 80% completed items is required.
Time Frame: 12 months after enrollment
Population: We imputed missing outcomes and covariates for TMLE analyses of this outcome. Therefore, all participants who enrolled in CISTO are included whether or not they completed that outcome. The mean and standard deviation for this outcome was calculated using only participants who completed this outcome (n = 238 and 143 for bladder-sparing therapy and radical cystectomy arms, respectively).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients who have selected bladder-sparing therapy | Patients who have selected radical cystectomy
Number analyzed (Participants) | 238 | 143
score on a scale | 47.1 (25.7) | 32.6 (20.1)
Statistical Analysis 1: Comparison: Patients who have selected bladder-sparing therapy vs Patients who have selected radical cystectomy; Test type: Other — We did not conduct a hypothesis test for this outcome. We presented an estimate of average treatment effect (ATE); TMLE = -11.9, 95% CI 2-sided [-14.7 to -9.0] — The ATE is interpreted as the causal mean difference in outcomes if all patients had been treated with RC versus having been treated with BST. A positive value indicates greater sexual health associated with radical cystectomy

8. Secondary Outcome: Patient Self-reported Sexual Health as Measured by the Bladder Cancer Index Sexual Summary Score
Description: as for outcome 7
Time Frame: 24 months after enrollment
Reporting Status: Not Posted

9. Secondary Outcome: Patient Self-reported Sexual Health as Measured by the Bladder Cancer Index Sexual Summary Score
Description: as for outcome 7
Time Frame: 60 months after enrollment
Reporting Status: Not Posted

10. Secondary Outcome: Patient Self-reported Bowel Health as Measured by the Bladder Cancer Index Bowel Summary Score
Description: The evaluation of the effect of treatment choice on patient-reported bowel health, as measured by the Bladder Cancer Index (BCI). The BCI consists of 36 items, with 4- or 5-point Likert response scales, covering 3 primary domains: urinary, bowel, and sexual. For each domain a summary score is constructed from the items used to calculate two subscale scores (function and bother). Scores are calculated by transforming item responses into a 0 to 100 scale and calculating the mean of the standardized items. Higher scores indicate better health status. To calculate a score, a minimum of 80% completed items is required.
Time Frame: 12 months after enrollment
Population: We imputed missing outcomes and covariates for TMLE analyses of this outcome. Therefore, all participants who enrolled in CISTO are included whether or not they completed that outcome. The mean and standard deviation for this outcome was calculated using only participants who completed this outcome (n = 293 and 166 for bladder-sparing therapy and radical cystectomy arms, respectively).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients who have selected bladder-sparing therapy | Patients who have selected radical cystectomy
Number analyzed (Participants) | 293 | 166
score on a scale | 80.1 (9.5) | 77.2 (10.8)
Statistical Analysis 1: Comparison: Patients who have selected bladder-sparing therapy vs Patients who have selected radical cystectomy; Test type: Other — We did not conduct a hypothesis test for this outcome. We presented an estimate of the average treatment effect (ATE); TMLE = -1.4, 95% CI 2-sided [-2.5 to -0.3] — The ATE is interpreted as the causal mean difference in outcomes if all patients had been treated with RC versus having been treated with BST. A negative value indicates worse bowel health associated with radical cystectomy

11. Secondary Outcome: Patient Self-reported Bowel Health as Measured by the Bladder Cancer Index Bowel Summary Score
Description: as for outcome 10
Time Frame: 24 months after enrollment
Reporting Status: Not Posted

12. Secondary Outcome: Patient Self-reported Bowel Health as Measured by the Bladder Cancer Index Bowel Summary Score
Description: as for outcome 10
Time Frame: 60 months after enrollment
Reporting Status: Not Posted

13. Secondary Outcome: Patient Self-reported Financial Distress as Measured by the Comprehensive Score for Financial Toxicity (COST)
Description: The evaluation of the effect of treatment choice on patient-reported financial distress, as measured by the Comprehensive Score for Financial Toxicity (COST). The COST questionnaire consists of 11 items, each scored on a 5-point Likert scale from zero to four. After reversing some items as indicated in the scoring manual (by reversing the sign on the original zero to four score and adding four), all item response scores are summed into a single financial toxicity score ranging from 0 to 44, with higher scores indicating greater financial wellbeing. Each subscale requires responses for at least 50% of the items in that subscale in order to be calculated. Item nonresponse is accounted for by substituting the mean of the completed items in the subscale.
Time Frame: 12 months after enrollment
Population: We imputed missing outcomes and covariates for TMLE analyses of this outcome. Therefore, all participants who enrolled in CISTO are included whether or not they completed that outcome. The mean and standard deviation for this outcome was calculated using only participants who completed this outcome (n = 288 and 167 for bladder-sparing therapy and radical cystectomy arms, respectively).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients who have selected bladder-sparing therapy | Patients who have selected radical cystectomy
Number analyzed (Participants) | 288 | 166
score on a scale | 30.4 (9.9) | 31.0 (9.4)
Statistical Analysis 1: Comparison: Patients who have selected bladder-sparing therapy vs Patients who have selected radical cystectomy; Test type: Other — We did not conduct a hypothesis test for this outcome. We presented an estimate of the average treatment effect (ATE); TMLE = 1.4, 95% CI 2-sided [0.2 to 2.6] — The ATE is interpreted as the causal mean difference in outcomes if all patients had been treated with RC versus having been treated with BST. A positive value indicates greater financial health associated with radical cystectomy

14. Secondary Outcome: Patient Self-reported Financial Distress as Measured by the Comprehensive Score for Financial Toxicity (COST)
Description: as for outcome 13
Time Frame: 24 months after enrollment
Reporting Status: Not Posted

15. Secondary Outcome: Patient Self-reported Financial Distress as Measured by the Comprehensive Score for Financial Toxicity (COST)
Description: as for outcome 13
Time Frame: 60 months after enrollment
Reporting Status: Not Posted

16. Secondary Outcome: Patient-reported Anxiety as Measured by the Patient Reported Outcome Measurement Information System (PROMIS) Short Form v1.0 - Anxiety 4a
Description: The evaluation of patient-reported anxiety, as measured by the Patient Reported Outcome Measurement Information System (PROMIS) Short Form v1.0 - Anxiety 4a. Scores range from 0 to 100, with higher scores indicating greater symptoms. Scores are normalized to a mean of 50 and standard deviation of 10.
Time Frame: 12 months after enrollment
Population: We imputed missing outcomes and covariates for TMLE analyses of this outcome. Therefore, all participants who enrolled in CISTO are included whether or not they completed that outcome. The mean and standard deviation for this outcome was calculated using only participants who completed this outcome (n = 294 and 169 for bladder-sparing therapy and radical cystectomy arms, respectively).
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Patients who have selected bladder-sparing therapy | Patients who have selected radical cystectomy
Number analyzed (Participants) | 294 | 169
T-score | 50.0 (8.9) | 48.8 (8.9)
Statistical Analysis 1: Comparison: Patients who have selected bladder-sparing therapy vs Patients who have selected radical cystectomy; Test type: Other — We did not conduct a hypothesis test for this outcome. We presented an estimate of the average treatment effect (ATE); TMLE = -2.4, 95% CI 2-sided [-3.1 to -1.6]; The ATE is interpreted as the causal mean difference in outcomes if all patients had been treated with RC versus having been treated with BST. A negative value indicates lower anxiety associated with radical cystectomy

17. Secondary Outcome: Patient-reported Anxiety as Measured by the Patient Reported Outcome Measurement Information System (PROMIS) Short Form v1.0 - Anxiety 4a
Description: as for outcome 16
Time Frame: 24 months after enrollment
Reporting Status: Not Posted

18. Secondary Outcome: Patient-reported Anxiety as Measured by the Patient Reported Outcome Measurement Information System (PROMIS) Short Form v1.0 - Anxiety 4a
Description: as for outcome 16
Time Frame: 60 months after enrollment
Reporting Status: Not Posted

19. Secondary Outcome: Patient-reported Depression as Measured by the Patient Reported Outcome Measurement Information System (PROMIS) Short Form v1.0 - Depression 4a
Description: The evaluation of patient-reported depression, as measured by the Patient Reported Outcome Measurement Information System (PROMIS) Short Form v1.0 - Depression 4a. Scores range from 0 to 100, with higher scores indicating greater symptoms. Scores are normalized to a mean of 50 and standard deviation of 10.
Time Frame: 12 months after enrollment
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Patients who have selected bladder-sparing therapy | Patients who have selected radical cystectomy
Number analyzed (Participants) | 294 | 169
T-score | 48.0 (8.3) | 48.0 (8.2)
Statistical Analysis 1: Comparison: Patients who have selected bladder-sparing therapy vs Patients who have selected radical cystectomy; Test type: Superiority — We did not conduct a hypothesis test for this outcome. We presented an estimate of the average treatment effect (ATE); TMLE = -1.0, 95% CI 2-sided [-1.8 to -0.3]; The ATE is interpreted as the causal mean difference in outcomes if all patients had been treated with RC versus having been treated with BST. A negative value indicates less depression associated with radical cystectomy

20. Secondary Outcome: Patient-reported Depression as Measured by the Patient Reported Outcome Measurement Information System (PROMIS) Short Form v1.0 - Depression 4a
Description: as for outcome 19
Time Frame: 24 months after enrollment
Reporting Status: Not Posted

21. Secondary Outcome: Patient-reported Depression as Measured by the Patient Reported Outcome Measurement Information System (PROMIS) Short Form v1.0 - Depression 4a
Description: as for outcome 19
Time Frame: 60 months after enrollment
Reporting Status: Not Posted

22. Secondary Outcome: Patient-reported Generic Quality of Life as Measured by the EuroQoL EQ-5D-5L
Description: The evaluation of patient-reported generic quality of life as measured by the EuroQoL EQ-5D-5L (EQ-5D). Scores range from 0 to 1, with higher scores indicating better health.
Time Frame: 12 months after enrollment
Population: We imputed missing outcomes and covariates for TMLE analyses of this outcome. Therefore, all participants who enrolled in CISTO are included whether or not they completed that outcome. The mean and standard deviation for this outcome was calculated using only participants who completed this outcome (n = 278 and 162 for bladder-sparing therapy and radical cystectomy arms, respectively).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients who have selected bladder-sparing therapy | Patients who have selected radical cystectomy
Number analyzed (Participants) | 278 | 162
score on a scale | 0.84 (0.14) | 0.86 (0.13)
Statistical Analysis 1: Comparison: Patients who have selected bladder-sparing therapy vs Patients who have selected radical cystectomy; Test type: Other — We did not conduct a hypothesis test for this outcome. We presented an estimate of the average treatment effect (ATE); TMLE = 0.03, 95% CI 2-sided [0.01 to 0.04]; The ATE is interpreted as the causal mean difference in outcomes if all patients had been treated with RC versus having been treated with BST. A positive value indicates greater quality of life associated with radical cystectomy

23. Secondary Outcome: Patient-reported Generic Quality of Life as Measured by the EuroQoL EQ-5D-5L
Description: as for outcome 22
Time Frame: 24 months after enrollment
Reporting Status: Not Posted

24. Secondary Outcome: Patient-reported Generic Quality of Life as Measured by the EuroQoL EQ-5D-5L
Description: as for outcome 22
Time Frame: 60 months after enrollment
Reporting Status: Not Posted

25. Secondary Outcome: Patient Recurrence-free Survival
Description: The evaluation of the effect of treatment choice on recurrence-free survival. Survival times were calculated from the date of diagnosis of recurrent high-grade non-muscle invasive bladder cancer to the event (recurrence or death). A recurrence was defined as any subsequent episode of high-grade bladder cancer in the bladder or elsewhere in the urinary tract (penile urethra, prostatic urethra, ureters, renal pelvis), either non-muscle or muscle invasive bladder cancer (for cystectomy arm this excludes any finding at cystectomy). Censoring occurred at the last electronic health record review or death.
Time Frame: 12 months after diagnosis of recurrent high-grade non-muscle invasive bladder cancer, up to 12 months post enrollment
Population: All participants who had an electronic health record review or death record at least 12 months after the diagnosis of recurrent high-grade non-muscle invasive bladder cancer. Survival times were calculated from the date of recurrence to the event (metastasis or death). Censoring occurred at the last electronic health record review or death.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients who have selected bladder-sparing therapy | Patients who have selected radical cystectomy
Number analyzed (Participants) | 356 | 192
Participants | 226 | 176
Statistical Analysis 1: Comparison: Patients who have selected bladder-sparing therapy vs Patients who have selected radical cystectomy; Test type: Other — We did not conduct a hypothesis test for this outcome; Risk Ratio (RR) = 1.45, 95% CI 2-sided [1.33 to 1.59] — Inverse probability weighted risk ratios calculated using quasi-Poisson regression. A weighted risk ratio > 1 implies that participants who choose RC have a greater chance of surviving without recurrence than those who choose BST

26. Secondary Outcome: Patient Recurrence-free Survival
Description: as for outcome 25
Time Frame: 24 months after diagnosis of recurrent high-grade non-muscle invasive bladder cancer
Reporting Status: Not Posted

27. Secondary Outcome: Patient Recurrence-free Survival
Description: as for outcome 25
Time Frame: 60 months after diagnosis of recurrent high-grade non-muscle invasive bladder cancer
Reporting Status: Not Posted

28. Secondary Outcome: Patient Metastasis-free Survival
Description: The evaluation of the effect of treatment choice on metastasis-free survival. Survival times were calculated from the date of diagnosis of recurrent high-grade non-muscle invasive bladder cancer to the event (metastatis or death). A metastasis was defined as metastasis to distant lymph/nodes organs (pathologic or radiologic diagnosis of M+ disease) (for cystectomy arm this includes findings at cystectomy). Censoring occurred at the last electronic health record review or death.
Time Frame: 12 months after diagnosis of recurrent high-grade non-muscle invasive bladder cancer, up to 12 months post enrollment
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Patients who have selected bladder-sparing therapy | Patients who have selected radical cystectomy
Number analyzed (Participants) | 349 | 192
Participants | 330 | 178
Statistical Analysis 1: Comparison: Patients who have selected bladder-sparing therapy vs Patients who have selected radical cystectomy; Test type: Other — We did not conduct a hypothesis test for this outcome; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.94 to 1.03] — Inverse probability weighted risk ratios calculated using quasi-Poisson regression. A weighted risk ratio < 1 implies that participants who choose RC have a lower chance of surviving without metastasis than those who choose BST

29. Secondary Outcome: Patient Metastasis-free Survival
Description: as for outcome 28
Time Frame: 24 months after diagnosis of recurrent high-grade non-muscle invasive bladder cancer
Reporting Status: Not Posted

30. Secondary Outcome: Patient Metastasis-free Survival
Description: as for outcome 28
Time Frame: 60 months after diagnosis of recurrent high-grade non-muscle invasive bladder cancer
Reporting Status: Not Posted

31. Secondary Outcome: Patient Progression-free Survival
Description: The evaluation of the effect of treatment choice on metastasis-free survival. Survival times were calculated from the date of diagnosis of recurrent high-grade non-muscle invasive bladder cancer to the event (metastatis or death). A progression was defined as any subsequent episode of muscle-invasive (T2-T4) disease in the bladder or elsewhere in the urinary tract AND/OR locoregional (true pelvic/common iliac) nodal disease (N+) AND/OR distant metastasis (M+) (for cystectomy arm this includes findings at cystectomy). Censoring occurred at the last electronic health record review or death.
Time Frame: 12 months after diagnosis of recurrent high-grade non-muscle invasive bladder cancer, up to 12 months post enrollment
Population: All participants who had an electronic health record review or death record at least 12 months after the diagnosis of recurrent high-grade non-muscle invasive bladder cancer. Survival times were calculated from the date of recurrence to the event (progression or death). Censoring occurred at the last electronic health record review or death.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients who have selected bladder-sparing therapy | Patients who have selected radical cystectomy
Number analyzed (Participants) | 349 | 194
Participants | 319 | 141
Statistical Analysis 1: Comparison: Patients who have selected bladder-sparing therapy vs Patients who have selected radical cystectomy; Test type: Other — We did not conduct a hypothesis test for this outcome; Risk Ratio (RR) = 0.80, 95% CI 2-sided [0.73 to 0.88] — Inverse probability weighted risk ratios calculated using quasi-Poisson regression. A weighted risk ratio < 1 implies that participants who choose RC have a lower chance of surviving without cancer progression than those who choose BST

32. Secondary Outcome: Patient Progression-free Survival
Description: as for outcome 31
Time Frame: 24 months after diagnosis of recurrent high-grade non-muscle invasive bladder cancer
Reporting Status: Not Posted

33. Secondary Outcome: Patient Progression-free Survival
Description: as for outcome 31
Time Frame: 60 months after diagnosis of recurrent high-grade non-muscle invasive bladder cancer
Reporting Status: Not Posted

34. Secondary Outcome: Patient Bladder Cancer-specific Survival
Description: The evaluation of the effect of treatment choice on bladder cancer-specific survival. Survival times were calculated from the date of diagnosis of recurrent high-grade non-muscle invasive bladder cancer to the event (death from bladder cancer). Censoring occurred at the last electronic health record review or date of death from bladder cancer.
Time Frame: 12 months after diagnosis of recurrent high-grade non-muscle invasive bladder cancer, up to 12 months post enrollment
Population: All participants who had an electronic health record review or death record at least 12 months after the diagnosis of recurrent high-grade non-muscle invasive bladder cancer. Survival times were calculated from the date of recurrence to the event (death from bladder cancer). Censoring occurred at the last electronic health record review or death from bladder cancer.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients who have selected bladder-sparing therapy | Patients who have selected radical cystectomy
Number analyzed (Participants) | 364 | 199
Participants | 359 | 192
Statistical Analysis 1: Comparison: Patients who have selected bladder-sparing therapy vs Patients who have selected radical cystectomy; Test type: Other — We did not conduct a hypothesis test for this outcome; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.96 to 1.01] — Inverse probability weighted risk ratios calculated using quasi-Poisson regression. A weighted risk ratio < 1 implies that participants who choose RC have a lower chance of surviving cancer than those who choose BST

35. Secondary Outcome: Patient Bladder Cancer-specific Survival
Description: as for outcome 34
Time Frame: 24 months after diagnosis of recurrent high-grade non-muscle invasive bladder cancer
Reporting Status: Not Posted

36. Secondary Outcome: Patient Bladder Cancer-specific Survival
Description: as for outcome 34
Time Frame: 60 months after diagnosis of recurrent high-grade non-muscle invasive bladder cancer
Reporting Status: Not Posted

37. Secondary Outcome: Patient Overall Survival
Description: The evaluation of the effect of treatment choice on overall survival. Survival times were calculated from the date of diagnosis of recurrent high-grade non-muscle invasive bladder cancer to the event (death). Censoring occurred at the last electronic health record review or date of death.
Time Frame: 12 months after diagnosis of recurrent high-grade non-muscle invasive bladder cancer, up to 12 months post enrollment
Population: All participants who had an electronic health record review or submitted a survey at least 12 months after the diagnosis of recurrent high-grade non-muscle invasive bladder cancer or had a death record at any time were included. Participants who did not have an electronic health record review or submit a survey at least 12 months after the diagnosis of recurrent high-grade non-muscle invasive bladder cancer and did not have a death record at any time were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients who have selected bladder-sparing therapy | Patients who have selected radical cystectomy
Number analyzed (Participants) | 364 | 199
Participants | 351 | 190
Statistical Analysis 1: Comparison: Patients who have selected bladder-sparing therapy vs Patients who have selected radical cystectomy; Test type: Superiority — Inverse probability weighted risk ratios calculated using quasi-Poisson regression; Risk Ratio (RR) = 0.89, 95% CI 2-sided [0.38 to 2.08] — A weighted risk ratio < 1 implies that participants who choose radical cystectomy have a lower chance of surviving than those who choose bladder-sparing therapy

38. Secondary Outcome: Patient Overall Survival
Description: as for outcome 37
Time Frame: 24 months after diagnosis of recurrent high-grade non-muscle invasive bladder cancer
Reporting Status: Not Posted

39. Secondary Outcome: Patient Overall Survival
Description: as for outcome 37
Time Frame: 60 months after diagnosis of recurrent high-grade non-muscle invasive bladder cancer
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Time frame for all-cause mortality is 12 months post enrollment to match participant flow. Time frame for all other adverse events is 12 months after diagnosis of recurrent high-grade non-muscle invasive bladder cancer, up to 12 months post enrollment.
Description: Adverse event reporting occurred systematically through regular investigator assessment and a standard questionnaire
Groups:
- Patients who have selected radical cystectomy: Patients with a diagnosis of recurrent high-grade NMIBC who have selected radical cystectomy (RC)
Arm/Group | Patients who have selected bladder-sparing therapy | Patients who have selected radical cystectomy
All-Cause Mortality (participants affected / at risk) | 19/371 | 11/199
Serious Adverse Events (participants affected / at risk) | 25/371 | 29/199
Other Adverse Events (participants affected / at risk) | 77/371 | 73/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients who have selected bladder-sparing therapy (N=371) | Patients who have selected radical cystectomy (N=199)
Abdominal infection (Infections and infestations) | 1 | 2
Lung infection (Infections and infestations) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Sepsis (Infections and infestations) | 3 | 3
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Postoperative hemorrhage (Surgical and medical procedures) | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Wound dehiscence (Surgical and medical procedures) | 0 | 2
(General disorders) | 18 | 22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patients who have selected bladder-sparing therapy (N=371) | Patients who have selected radical cystectomy (N=199)
Hematuria (Renal and urinary disorders) | 32 | 6
Urinary tract infection (UTI) (Renal and urinary disorders) | 41 | 32
Anemia (Blood and lymphatic system disorders) | 12 | 40
Nausea (Gastrointestinal disorders) | 13 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/26/NCT03933826/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT03933826/SAP_001.pdf